CLINICAL TRIAL: NCT06184035
Title: Ph I/IIa Escalation/Expansion FIH, Open, Multi Center, Single Arm Study Evaluating Safety, Dosimetry and Early Efficacy of 177Lu-SN201 in Progressive/Treatment-refractory, Locally Advanced, Unresectable Metastatic or Recurrent Solid Tumors
Brief Title: A Dose Escalation and Expansion Study of [177Lu]Lu-SN201 in Participants With Advanced Cancer
Acronym: Tumorad
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spago Nanomedical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tumorad-01
Record Dates: First submitted 2023-12-06; First posted 2023-12-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor; Metastatic Cancer; Unresectable Solid Tumor; Recurrent Solid Tumor; Locally Advanced Solid Tumor; Refractory Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I/IIa Dose escalation and dose expansion (Experimental): Participants will initially receive 1 cycle of [177Lu]Lu-SN201 via slow intravenous infusion and progress to up to 3 cycles, provided retreatment criteria are met before the start of each cycle, occurring every 6 weeks (with an allowable window to delay each cycle by +3 weeks per retreatment criteria).
  Dose escalation: The study will evaluate up to 5 dose levels of [177Lu]Lu-SN201 (A1=10 MBq/kg, A2=25 MBq/kg, A=50 MBq/kg, A4= <33% of A3, A5= <33% of A4). Additional dose levels may be explored until MTD/RP2D is identified. Up to 9 participants may be enrolled at any pre-specified dose level shown to be tolerated for confirmation of MTD and/or RP2D.
  Dose expansion: Once the MTD/RP2D has been defined, an expansion phase consisting of multiple tumor types, each with up to 20 participants, will be enrolled to further characterize the safety, tolerability, and assess preliminary efficacy of [177Lu]Lu-SN201 at the RP2D and/or MTD identified in Phase I.
  Interventions: Drug: [177Lu]Lu-SN201

INTERVENTIONS:
Drug: [177Lu]Lu-SN201 — Intravenous infusion
  Other Names: Tumorad

SUMMARY:
The purpose of this first-in-human (FIH) study is to determine the maximum tolerated dose (MTD) and to characterize the safety, tolerability, PK, and dosimetry profile of [177Lu]Lu-SN201 in adult participants with advanced solid tumors who have no standard of care treatment options.

[177Lu]Lu-SN201 is a radiolabeled, nanomedical investigational medicinal product (IMP) whose mechanism of delivery is based on the Enhanced Permeability and Retention (EPR) effect.

DETAILED DESCRIPTION:
Eligible participants will receive [177Lu]Lu-SN201 via slow intravenous infusion on Cycle 1 Day 1. Participants will initially receive one cycle of treatment and will progress to a 2nd and 3rd cycle of treatment, provided retreatment criteria are met before the start of each cycle. The dosing schedule visit frequency will be every 6 weeks (with an allowable window to delay each cycle by +3 weeks per retreatment criteria), each participant may receive up to 3 cycles, with the treatment duration up to 22 weeks. A total of 3 treatment cycles will be given unless the participant meets early discontinuation criteria. For Cycle 1, an overnight hospitalization for standard-of-care observation following Day 1 clinic assessments to Day 2 is mandatory for all participants receiving Cycle 1.

Whole-body planar imaging, and single photon emission computed tomography (SPECT)/computed tomography (CT) will be performed post-administration of [177Lu]Lu-SN201 to assess biodistribution and dosimetry. CT or magnetic resonance imaging (MRI) will be used to assess the response of the disease to treatment using Response Evaluation Criteria (RECIST v1.1).

The general procedures for participants in Phase I and Phase IIa are summarized below:

* Baseline values are defined as the last collected value prior to the start of infusion.
* Continual assessment of adverse events (AEs) and concomitant medication usage will be conducted.
* Whole-body planar on Day 1, Day 2, Day 4, and Day 8 and SPECT/CT on Day 2, Day 4 and Day 8 will be used for biodistribution and dosimetry evaluation of all participants. If dosimetry has been met by previous participants at each dose level, the DMC may partly or fully exclude the requirement for dosimetry procedures in remaining participants at this dose level.
* For participants that will continue to treatment Cycle 2 or 3, eligibility assessment and IMP procurement will take place within the coming 17 days.

ELIGIBILITY:
Inclusion criteria:

1. Male or female participants ≥ 18 years of age on the day of signing informed consent.
2. Histologically or cytologically documented, recurrent, locally advanced, or metastatic solid malignancy that has failed at least one prior systemic standard therapy, or for which standard therapy is not appropriate, or for which no standard therapy exists.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. Life expectancy ≥ 3 months.
5. Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements, to be conducted within 28 days before the start of the study IMP administration:

   1. Hemoglobin ≥ 9.0 g/dL (transfusions are allowed).
   2. Absolute neutrophil count (ANC) ≥ 1500/mm3.
   3. Platelet count ≥ 100,000 mm3.
   4. Total bilirubin ≤ 2.5 x upper limit of normal (ULN) (in participants with liver metastases ≤ 5 ULN).
   5. Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 5 x ULN.
6. On a stable dose of anti-coagulation therapy will be allowed to participate if they have no sign of bleeding or clotting and prothrombin/international normalized ratio and partial thromboplastin time (PT/INR and PTT, respectively) test results are compatible with the acceptable benefit-risk ratio at the Investigator's discretion.
7. Serum creatinine ≤ 1.5 x ULN and estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m2 (per local values).
8. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   1. Male participants must agree to use a highly effective method of birth control as defined in ICH M3(R2) starting with the first dose of study medication through 120 days after the last dose of study medication.
   2. Female participants of childbearing potential* must have a negative pregnancy test documented at Screening and Baseline and be willing to use a highly effective method of contraception** or practice abstinence starting from ICF signature through to 120 days after the last dose of study medication.

      * A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy or bilateral oophorectomy, or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., had had menses at any time in the preceding 24 consecutive months).

        * Effective contraception is defined as contraceptive methods with a failure rate of < 1% to prevent pregnancy (combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system).
9. Written informed consent to study participation.
10. Be able to understand and comply with the requirements of the study, as judged by the Investigator.
11. Phase I: At least one lesion as per RECIST v1.1.
12. Phase IIa: At least one measurable lesion as per RECIST v1.1.

Exclusion criteria:

1. Unstable systemic disease (including but not limited to active infection, hepatic, renal, or metabolic disease).
2. Clinically significant cardiac disease including any of the following:

   1. Congestive heart failure requiring treatment (New York Heart Association Grade ≥ 2).
   2. LVEF of < 50%, as determined by MUGA or ECHO.
   3. Uncontrolled hypertension, defined as persistent systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy.
   4. History or presence of clinically significant ventricular arrhythmias or atrial fibrillation.
   5. Clinically significant resting bradycardia.
   6. Unstable angina pectoris ≤ 3 months before the start of study treatment.
   7. Acute myocardial infarction ≤ 3 months before the start of study treatment.
   8. Mean triplicate QT interval corrected for heart rate using Fridericia's formula (QTcF) value > 480 msec (as specified in Section 10.5).
3. Known hypersensitivity to pegylated drugs or vaccines (e.g., covid-19 vaccines).
4. Concurrent or active solid or hematologic malignancy within the last 2 years with a distinct primary site or histology from the cancer being evaluated in this study except for the following cancer types: cervical cancer in situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis).
5. Infections not responding to therapy or active clinically serious infections.
6. Known human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection requiring treatment. Participants with chronic HBV or HCV infection are eligible at the Investigator's discretion provided that the disease is stable and sufficiently controlled under treatment.

   NB: Participants with CNS metastases may be included after discussion with Sponsor, except for the sentinel participants.
7. Chemotherapy, experimental cancer therapy, biologic therapy, or immunotherapy within 2 weeks (or 5 half-lives, whatever is shortest) before the start of the study IMP administration.
8. Palliative radiotherapy completed less than 2 weeks before the start of the study IMP administration will be allowed as long as no more than 10% of the participant's bone marrow was irradiated.
9. Not recovered to Grade 1 from any prior anti-cancer therapy, excluding alopecia.
10. Previous high-dose chemotherapy needing hemopoietin-stem-cell-rescue.
11. Major surgery, open biopsy, or significant trauma within 4 weeks before the start of study treatment.
12. A psychiatric or functional disorder that prevents participants from providing informed consent or following protocol instructions.
13. A participant that has a condition or is in a situation, in the Investigator's opinion may put the individual at significant risk, may confound the study results, or may interfere significantly with their participation in the study.
14. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks or 5 half-lives of the agent, whichever is the shortest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I/IIa: Frequency and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 48 months
  Clinically significant safety laboratory results will be graded by NCI CTCAE v5.0. AEs (including physical examination, vital signs, ECG, and safety lab findings), related AEs, DLTs, SAEs, and related SAEs, AEs with NCI CTCAE Grades ≥ 3, AEs leading to premature discontinuation, interruptions, duration of interruptions and discontinuation of IRP will be analyzed descriptively utilizing corresponding Medical Dictionary for Regulatory Activities System Organ Classes and Preferred Terms. NCI CTCAE v5.0 toxicity grades will be utilized for classifying severity.
  Continual assessment of adverse events (AEs) and concomitant medication usage will be conducted.
Phase I/IIa: Incidence of Dose-Limiting Toxicity (DLT) during the first cycle of treatment. | 48 months
  DLTs are defined as:
  * Any Grade ≥ 3 AEs of any etiology that are clinically significant and last > 7 days except:
    * Nausea, vomiting, or diarrhea will be considered a DLT only if it persists at Grade ≥ 3 for > 3 days despite adequate supportive care measures. At the Investigator's discretion, participants who experience nausea, vomiting, or diarrhea after receiving IMP may receive antiemetic or anti-diarrheal medication before subsequent doses of IMP.
    * Isolated laboratory abnormalities Grade ≥ 3 (not present at Baseline) that are not considered to be significant by the Investigator and are resolved to at least Grade 1 within 7 days without clinical sequelae or need for therapeutic intervention.
  * Any other toxicity occurring at any time during the study that in the view of the participating Investigators and the Medical Monitor represents a clinically significant hazard to the participant.
  DLTs will be confirmed by the DMC.
Phase I: Dose escalation to identify RP2D and/or MTD dose | 24 months
  RP2D and/or MTD will be based on the DLT rate. Dose escalation will follow BOIN design, directed by the DLT rate (the current number of participants with DLT divided by the current number of participants in the cohort).
  The study will evaluate up to 5 dose levels of [177Lu]Lu-SN201, however additional dose levels may be explored until MTD/RP2D is identified. If the starting dose is not tolerated, a lower dose may be evaluated based on toxicity, safety, pharmacokinetics, and dosimetry data as determined by the DMC.
Phase IIa: Clinical benefit in solid tumor subgroups at RP2D and/or MTD | 24 months
  Clinical benefit according to RECIST v1.1 of [177Lu]Lu-SN201, as defined by post-treatment tumor response and serum levels of applicable tumor markers, compared to baseline (last collected value/measurement before the start of treatment)

SECONDARY OUTCOMES:
Phase I/IIa: Measure peak plasma [177Lu]Lu-SN201 activity concentration (Cmax) | 48 months
  Characterize the pharmacokinetic Peak plasma concentration (Cmax) of the [177Lu]Lu-SN201 activity concentration over time
Phase I/IIa: Measure plasma half-life of the [177Lu]Lu-SN201 activity | 48 months
  Characterize the pharmacokinetic half-life of the [177Lu]Lu-SN201 activity concentration over time in plasma
Phase I/IIa: Measure the area under the plasma concentration versus time curve (AUC) of [177Lu]Lu-SN201 activity | 48 months
  Characterize the pharmacokinetic area under the curve vs time curve of the [177Lu]Lu-SN201 activity concentration in plasma over time
Phase I/IIa: Evaluation of clinical dosimetry | 48 months
  To evaluate clinical dosimetry with whole-body planar and SPECT/CT imaging modalities to asses percentage injected dose of activity concentration and distribution of [177Lu]Lu-SN201 in tumor and organs.
Phase IIa: Evaluation of clinical benefit based on disease control rates (DCR) | 12 months
  To evaluate clinical benefit based disease control rates (DCR) according to RECIST v1.1;
  * Overall Response Rate (ORR).
  * Duration of response (DoR).
  * Progression-free survival (PFS).
  * Overall survival (OS).

OTHER OUTCOMES:
Phase I: Evaluation of clinical benefit based on disease control rates (DCR) | 12 months
  To evaluate clinical benefit based disease control rates (DCR) according to RECIST v1.1;
  * Overall Response Rate (ORR).
  * Duration of response (DoR).
  * Progression-free survival (PFS).
  * Overall survival (OS).
Phase I: Characterization of early signs of efficacy in tumor-type subgroups | 24 months
  Up to 3 subgroups will be selected for the Phase IIa part of the study, based on emerging data on early signs of efficacy, and discussions with Clinical Investigators and Sponsor representatives.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Taubman, Principal Investigator — St Vincent Hospital Melbourne
Locations (2):
- Australia (2):
  - Cancer Research South Adelaide, Adelaide, South Australia
  - St Vincent Hospital Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No